CLINICAL TRIAL: NCT02976064
Title: Protocol for Implementation of Collaborative Self-management Services to Promote Physical Activity
Brief Title: Implementation of Collaborative Self-management Services to Promote Physical Activity
Acronym: NEXTCARE-PA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Badalona Serveis Assistencials (Other); Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Josep Roca, Consultor senior, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NEXTCARE-PA
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chronic Disease
Keywords: physical activity; lifestyle; adaptive case management; telemedicine; integrated care; collaborative self-management
MeSH Terms: conditions — Chronic Disease; Motor Activity | interventions — Preoperative Exercise; Rehabilitation; Primary Health Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PreHab_Intervention (Experimental): Experimental group of the prehabilitation trial
  Interventions: Behavioral: PreHabilitation
- PreHab_Control (No Intervention): Control group of the prehabilitation trial
- Chronic patients_Intervention (Experimental): Experimental group of the Rehabilitation in chronic stable patients in primary care trial
  Interventions: Behavioral: Rehabilitation in chronic stable patients in primary care
- Chronic patients_Control (No Intervention): Control group of the Rehabilitation in chronic stable patients in primary care trial
- Citizens & mild disease_Intervention (Experimental): Experimental group of the Rehabilitation in mild chronic patients and citizens at risk trial
  Interventions: Behavioral: Rehabilitation in mild chronic patients and citizens at risk
- Citizens & mild disease_Control (No Intervention): Control group of the Rehabilitation in mild chronic patients and citizens at risk trial

INTERVENTIONS:
Behavioral: PreHabilitation — 1. Case identification: Candidates fulfilling the inclusion criteria will be identified by the anesthesiologist.
  2. Case evaluation: Candidates will be assessed to identify the overall needs and perform a baseline evaluation.
  3. Personalized Work plan definition: Personalization of the plan involves a calendar and planning of face to face visits and remote contacts; intensity of the supervised exercise training program; threshold of steps per day; nutritional intervention; psychological intervention; and integration of the intervention into the overall work plan.
  4. Work plan execution & 5-Follow-up+event handling: Involve the follow-up tasks, including non-scheduled interactions through the personal health folder (PHF)
  6-Discharge: Patient will be discharged from prehabilitation and moved to rehabilitation.
  Arms: PreHab_Intervention
Behavioral: Rehabilitation in chronic stable patients in primary care — 1. Case identification: Candidates fulfilling the inclusion criteria will be identified by the general practitioner.
  2. Case evaluation: The primary care team will characterize the candidates, covering: i) patient requirements defining the work plan; ii) aerobic capacity and physical activity; iii) identification of factors modulating adherence.
  3. Personalized work plan definition: The community-based intervention will include reassessment of the patient's work plan aiming at optimization of both pharmacological and non-pharmacological therapies. Consist of a motivational interview and a physical activity (PA) intervention (6-month duration) based on supervised endurance training, promotion of PA and empowerment for self-management using the PHF.
  4. Work plan execution & 5-Follow-up+event handling: The ICT-support will facilitate the program follow up.
  6-Discharge: The patient will be discharged or moved to the PA service addressed to citizens at risk & patients with mild disease.
  Arms: Chronic patients_Intervention
Behavioral: Rehabilitation in mild chronic patients and citizens at risk — 1. Case identification: Candidates fulfilling the inclusion criteria will be identified by the GP.
  2. Case evaluation: i) patient requirements defining the work plan; ii) aerobic capacity and PA; iii) identification of factors modulating adherence.
  3. Personalized work plan definition: i) motivational interview; ii) training for the use of the PHF for self-management; and iii) assign one case manager for off-line remote surveillance. The following optional modules are envisaged: i) basic service (above); ii) endurance training programs; iii) community physical activity group sessions; and/or, iv) upgraded PA program including sensors and close off-line supervision.
  4. Work plan execution & 5-Follow-up+event handling: The ICT-support will facilitate the program follow up.
  6-Discharge: The basic version of the promotion of PA program is conceived for a timeless duration. However, the different modules included in the service portfolio will have specific agendas and associated costs.
  Arms: Citizens & mild disease_Intervention

SUMMARY:
Background: The growing awareness on the health burden generated by insufficient levels of physical activity has prompted the interest for deploying community-based initiatives aiming at fostering active healthy living. It is of note, however, that, to our knowledge, none of the interventions evaluated so far have reached large scale adoption. The current protocol relies on the general hypothesis that properly tailored self-management programs, fully integrated in the patient's action plan with remote off-line professional support, may induce sustained behavioral changes resulting in exercise health behavior. Accordingly, the current manuscript addresses those unmet requirements, namely: i) Workflow design of the PA services engaging both patients and health professionals; ii) Enhanced information and communication technologies (ICT)-support; iii) Evaluation strategies including structured indicators; and, iv) Implementation of innovative business models. The main outcome of the current protocol will be a roadmap for large scale deployment and assessment of novel collaborative self-management PA services in the region of Catalonia (7.5 million citizens).

Methods: The protocol has been designed as part of the regional deployment of integrated care services in Catalonia (2016-2020). It has been conceived has a two-year (2017-2018) test bed period.

Aims: The protocol uses a population-health approach to addresses the four aims: i) Prehabilitation for high risk candidates to major surgery; ii) Community-based rehabilitation for clinical stable chronic patients with moderate to severe disease; and, iii) Promotion of physical activity and healthy lifestyles for citizens at risk and patients with mild disease.

ELIGIBILITY:
Inclusion Criteria:

Arms 1 & 2:

* Candidates to major elective surgical procedures in the following specialties: abdominal, gynecology, cardiovascular, urology and thoracic
* Patients presenting high surgical risk because they are they are aged > 70 years and/or show an American Society of Anesthesiologist (ASA) score of III/IV
* A tentative surgical schedule allowing for at least 4 weeks for the pre-habilitation intervention.

Arms 3 & 4:

* Patients suffering one or more targeted chronic conditions (cardiovascular diseases, chronic obstructive pulmonary disease and type 2 diabetes mellitus)
* Moderate-to-severe disease (main disorder)
* High user of healthcare resources assessed by history of past hospital-related events (admissions and/or emergency room visits).

Arms 5 & 6:

* Citizens at risk for chronic conditions and patients showing mild target disease(s) recruited through advertisements, primary care centers or pharmacy offices.

Exclusion Criteria:

Arms 1 & 2:

* Emergency surgery
* Unstable cardiac or respiratory disease
* Locomotor limitations precluding the practice of exercise
* Cognitive deterioration impeding the adherence to the program.

Arms 3-6:

* Unstable cardiovascular or respiratory disorders
* Locomotor limitations precluding the practice of exercise
* Cognitive deterioration impeding the adherence to the program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications during hospitalization | Postoperative hospitalization period (up to 90 days)
  Primary outcome for arms 1 & 2 - Percentage of patients suffering postoperative complications during hospitalization
Determinants of adoption of the PA service | Life-span of the project (12 months)
  Primary outcome for arms 3 & 4
Changes in Health-related quality of life | Baseline - Six months - 12 months
  Primary outcome for arms 5 & 6 - Short-form 36 survey

SECONDARY OUTCOMES:
Changes in Aerobic capacity | Baseline - Six months - 12 months
  Six-minute walking test
Hospital length of stay | Postoperative hospitalization period (up to 90 days)
  Days of hospital stay
Intensive care unit length of stay | Postoperative hospitalization period (up to 90 days)
  Days of ICU stay
Changes in Physical activity | Baseline - Six months - 12 months
  Accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Josep Roca, Prof, Principal Investigator — Hospital Clinic de Barcelona - IDIBAPS - University of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barberan-Garcia A, Gimeno-Santos E, Blanco I, Cano I, Martinez-Palli G, Burgos F, Miralles F, Coca M, Murillo S, Sanz M, Steblin A, Ubre M, Benavent J, Vidal J, Sitges M, Roca J. Protocol for regional implementation of collaborative self-management services to promote physical activity. BMC Health Serv Res. 2018 Jul 17;18(1):560. doi: 10.1186/s12913-018-3363-8. PMID 30016944